CLINICAL TRIAL: NCT00493532
Title: An Open Label Study to Evaluate the Effect on Bone Mineral Density, and the Safety, of Quarterly Intravenous Bonviva in Patients With Post-menopausal Osteoporosis.
Brief Title: A Study of Quarterly Intravenous Bonviva (Ibandronate) in Women With Post-Menopausal Osteoporosis.
Status: No longer available | Type: Expanded Access
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML20882
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 3mg iv every 3 months

SUMMARY:
This single arm study will assess the efficacy and safety of quarterly intravenous Bonviva in women with post-menopausal osteoporosis. All patients will receive Bonviva 3mg i.v. every 3 months. The anticipated time on study treatment is 3-12 months, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women with osteoporosis;
* <=80 years of age;
* naive to oral bisphosphonates, or have discontinued daily and/or weekly bisphosphonate treatment for >1 year.

Exclusion Criteria:

* metabolic bone disease other than post-menopausal osteoporosis;
* treatment with other drugs affecting bone metabolism within last 6 months;
* previous or current malignant disease (except for adequately treated cancer in situ of the cervix, or basal or squamous cell skin cancer).

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Taiwan (7):
  - Chai Yi
  - Changhua
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District